CLINICAL TRIAL: NCT04163432
Title: A Randomized, Phase II Study of Staggered, Chemo-Immunotherapy With Durvalumab, MEDI4736 Pemetrexed and Carboplatin (PC) for Metastatic Non-Squamous NSCLC
Brief Title: Staggered, Chemo-Immunotherapy With Durvalumab, MEDI4736 Pemetrexed & Carboplatin (PC) for Metastatic Non-Squamous NSCLC
Acronym: STAGGER
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HCI127115
Record Dates: First submitted 2019-11-04; First posted 2019-11-14 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Non-Small Cell Lung Cancer Metastatic
MeSH Terms: interventions — durvalumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Intervention Model Description: Phase II, open label, randomized study of durvalumab in combination with pemetrexed and carboplatin in eligible adult patients with locally advanced or metastatic non-small cell lung cancer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Chemo-Immuno (Experimental): ArmA receives chemotherapy on D1 and immunotherapy on D8 of a 28-day cycle for the first 2cycles. After the first 2cycles, patients on Arm A and Arm B will be administered chemotherapy and immunotherapy on D1 of a 21day cycle for cycles 3 and 4. After 4cycles of chemo-immunotherapy, patients receive maintenance therapy with durvalumab and pemetrexed until treatment discontinuation. Maintenance therapy is administered on D1 of a 21day cycle.
  Interventions: Drug: Durvalumab; Drug: Pemetrexed; Drug: Carboplatin
- Arm B: Immuno-Chemo (Experimental): ArmB receives immunotherapy on D1 and chemotherapy on D8 of a 28-day cycle for the first 2cycles. After the first 2cycles, patients on Arm A and Arm B will be administered chemotherapy and immunotherapy on D1 of a 21day cycle for cycles 3 and 4. After 4cycles of chemo-immunotherapy, patients receive maintenance therapy with durvalumab and pemetrexed until treatment discontinuation. Maintenance therapy is administered on D1 of a 21day cycle.
  Interventions: Drug: Durvalumab; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Durvalumab — Durvalumab is administered at a dose of 1500mg for patients who weigh >30 kg. If weight falls to ≤ 30 kg, weight-based dosing at 20mg/kg will be a utilized
  Other Names: Imfinzi
Drug: Pemetrexed — Pemetrexed dosing is adjusted for kidney function. Pemetrexed is dosed at 500mg/m2 for patients with a creatinine clearance ≥ 45 mL/min (by Cockcroft-Gault formula). If creatinine clearance is < 45 mL/min, pemetrexed is dosed at 400 mg/m2.
  Other Names: Alimta
Drug: Carboplatin — Carboplatin dosing is adjusted for kidney function.The total dose (in mg) of carboplatin will be calculated using the Calvert Formula utilizing a target AUC of 5 and a patient's GFR in mL/min.

SUMMARY:
This is a Phase II, open label, randomized study of durvalumab in combination with pemetrexed and carboplatin in eligible adult patients with locally advanced or metastatic non-small cell lung cancer. The study will focus on the efficacy of two alternative staggered dosing regimens.

DETAILED DESCRIPTION:
This trial will evaluated two different schedules of concurrent chemoimmunotherapy while simultaneously measuring immune activation, immune resistance and host factors. Both arms will consist of concurrent chemoimmunotherapy with durvalumab, pemetrexed and carboplatin, but in arm 1 the chemotherapy will precede the immunotherapy by a week and in arm 2 the immunotherapy will precede the chemotherapy by a week. Staggering these therapies still allows concurrent administration while allowing some degree of temporal isolation to better understand the contributions by chemotherapy and immunotherapy in this setting. Host and laboratory factors will be measured during treatment. We hypothesize that staggered dosing of immunotherapy in combination with chemotherapy can improve clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged ≥ 18 years.
* Histologically or cytologically confirmed lung cancer.
* Metastatic non-squamous non-small cell lung cancer.
* Body weight >30kg
* Patient has measurable disease as defined by RECIST 1.1 as assessed by either CT or MRI.
* Chemoimmunotherapy naïve (including durvalumab).
* ECOG Performance Status ≤ 2. --Note: If performance status = 2, ensure that there is a slot available prior to registration as only 20 PS = 2 patients will be enrolled on the protocol.
* Must have a life expectancy of at least 12 weeks.
* Adequate organ function as defined as:

  * Hematologic:

    * White blood cell count > 2.0 g/dL
    * Platelet count ≥ 100,000/mm3
    * Hemoglobin ≥ 9 g/dL
    * Absolute neutrophil count (ANC) ≥ 1,500/mm3
  * Hepatic:

    ---Total Bilirubin ≤ 1.5 x institutional upper limit of normal (ULN)

    ---Except for patients with Gilbert's syndrome.

    ---AST(SGOT)/ALT(SGPT) ≤ 2.5 × institutional ULN or ≤ 5 × institutional ULN if liver metastases are present
  * Renal:

    * eGFR ≥ 30 mL/min/1.73m2 or creatinine clearance ≥ 30 mL/min by Cockcroft-Gault:
    * Males: ((140-age)×weight[kg])/(serum creatinine [mg/dL]×72)
    * Females: (((140-age)×weight[kg])/(serum creatinine [mg/dL]×72))×0.85
* FOR PATIENTS ENROLLED PRIOR TO AMENDMENT V18MAR2024: Concurrent enrollment in the study, "Rethinking Measurement of Performance Status in Cancer Patients," IRB 112529 or the patient declined participation.
* FOR PATIENTS ENROLLED PRIOR TO AMENDMENT V18MAR2024: Concurrent enrollment in the study, "An Observational Study Assessing the Clinical Effectiveness of the VeriStrat® Test and Validating Immunotherapy Tests in Subjects with Non-Small Cell Lung Cancer," IRB 100314 or the patient has declined participation.
* Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

  --Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).

  --Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
* Highly effective contraception for both male subjects with partners of childbearing potential and female subjects of childbearing potential throughout the study and for at least 90 days after the last dose of study therapy.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.

Exclusion Criteria:

* ALK or EGFR non-squamous non-small cell lung cancer.
* Prior radiation therapy within 2 weeks prior to cycle one day one.

  -Exception: Prior palliative radiotherapy is permitted, provided it has been completed at least 2 days prior to study enrollment and no clinically significant toxicities are expected.
* Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP.

  -Note: Local surgery of isolated lesions for palliative intent is acceptable.
* History of allogenic organ transplantation.
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis,uveitis, etc]). The following are exceptions to this criterion:

  * Patients with vitiligo or alopecia
  * Patients with endocrine disorders with controlled disease on hormone replacement therapy (e.g. adrenal, thyroid, or pituitary replacement therapy)
  * Any chronic skin condition that does not require systemic therapy
  * Patients without active disease in the last 5 years may be included but only after consultation with the principal investigator
  * Patients with celiac disease controlled by diet alone
* Current or prior use of immunosuppressive medication within 14 days of cycle one day one, EXCEPT for the following permitted steroids:

  * Intranasal, inhaled, topical steroids, eye drops or local steroid injection (eg,intra-articular injection);
  * Systemic corticosteroids at physiologic doses ≤ 10mg/day of prednisone or equivalent;
  * Steroids as premedication for hypersensitivity reactions (eg, computed tomography (CT) scan premedication).
  * Other immunosuppressive agents which, in the opinion of the investigator, are not expected to significantly impact study participation or the mechanism of action of the study therapy.
* History of active primary immunodeficiency
* Diagnosis of any other malignancy within 2 years prior to study enrollment, except for adequately treated basal cell or squamous cell skin cancer, carcinoma in situ of the breast, bladder or of the cervix, and low-grade (Gleason 6 or below) prostate cancer on surveillance with no plans for treatment intervention (eg, surgery, radiation, or castration) or prostate cancer that has been adequately treated with prostatectomy or radiotherapy and currently with no evidence of disease or symptoms is allowed.
* Uncontrolled CNS metastases; subjects with previously treated brain metastases will be allowed if the brain metastases have been treated, toxicities have resolved to grade 1 or baseline and steroids are no longer required.

  --Patients with asymptomatic brain metastasis are allowed if previous steroid treatment was discontinued for 5 half-lives.
* History of leptomeningeal carcinomatosis
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
* Known HIV infection that is not well controlled. All of the following criteria are required to define an HIV infection that is well controlled: undetectable viral RNA load 12 months, CD4+ count of ≥ 350 cells/uL, no history of AIDS-defining opportunistic infection within the past 12 months, and stable for at least 1 month on the same anti HIV medications.
* Active tuberculosis infection (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice).
* Known active hepatitis infection, positive hepatitis C virus (HCV) antibody, hepatitis B virus (HBV) surface antigen (HBsAg) or HBV core antibody (anti-HBc), at screening. Participants with a past or resolved HBV infection (defined as the presence of anti HBc and absence of HBsAg) are eligible. Participants positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Participants co-infected with HBV and HCV, or co-infected with HBV and HDV, namely: HBV positive (presence of HBsAg and/or anti HBcAb with detectable HBV DNA); AND

  1. HCV positive (presence of anti-HCV antibodies); OR
  2. HDV positive (presence of anti-HDV antibodies).
* Vaccination with a live vaccine within 30 days of cycle one day one and while on trial is prohibited except for administration of inactivated vaccines.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy
* Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies, cisplatin, other platinum-containing compounds, or mannitol. (NCI CTCAE v5.0 Grade ≥ 3).
* Subjects taking prohibited medications as described in Section 6.5.2. A washout period of prohibited medications for a period of at least 5 half-lives or as clinically indicated should occur prior to the start of treatment.
* Participation in another clinical study with an investigational product during the last 2 weeks.
* Concurrent enrollment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.

  * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
* Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at approximately 5 minutes apart).
* Patients who have received prior anti-PD-1, anti PD-L1 or anti CTLA-4.
* Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
* All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
* Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy.

NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.

*Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2020-06-16 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of clinical benefit | up to 5 years
  Described using RECIST 1.1 response criteria.

SECONDARY OUTCOMES:
Incidence of adverse events | up to 5 years
  Adverse events (AEs) and serious adverse events (SAEs) will be collected and assessed by CTCAE, v5.0 for assessment of safety and feasibility.
Objective response rate (ORR) | up to 5 years
  Assessed using RECIST 1.1
Progression free survival (PFS) | up to 5 years
  Assessed as the time between trial initiation and documented progression or radiographic imaging.
Overall survival (OS) | up to 5 years
  assessed as the time from trial initiation until death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Gumbleton, MD, Principal Investigator — Huntsman Cancer Institute
Locations (1):
- Huntsman Cancer Institute at University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No